CLINICAL TRIAL: NCT00292344
Title: Rifaximin in Standard Three-Day Dosing With and Without the Antimotility Drug, Loperamide, in the Treatment of Travelers' Diarrhea
Brief Title: Rifaximin, Loperamide and the Combination to Treat Travelers' Diarrhea
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: TRA-04-01
Record Dates: First submitted 2006-02-13; First posted 2006-02-15 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2006-02

CONDITIONS: Travelers' Diarrhea
Keywords: Travelers' diarrhea; rifaximin; loperamide; enterotoxigenic E. coli
MeSH Terms: interventions — Rifaximin; Loperamide

INTERVENTIONS:
Drug: Rifaximin and loperamide

SUMMARY:
Most cases of travelers' diarrhea are caused by bacterial pathogens which respond slowly to antibiotic treatment.The study was designed to determine the value of rapidly acting loperamide (imodium) combined with curative dose of the poorly absorbed rifaximin in travelers' diarreha treatment.

DETAILED DESCRIPTION:
During short-term study, adult U.S. students in Mexico (n = 310) with acute diarrhea (≥ 3 unformed stools with enteric symptoms) were enrolled in a double-blind, randomized trial wherein they were given rifaximin 200 mg three times a day for 3 days (R) (n = 102), loperamide 4 mg initially followed by 2 mg after each unformed stool not to exceed 8 mg/day for 2 days (L) (n = 104) or both drugs in the same dosage schedule (L/R) (n = 104). The major outcome parameter was time from initiation of therapy until passage of the last unformed stool before becoming well (TLUS).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include: IRB approval; signing of a consent form;18 years of age or older, providing of an unformed pre-treatment stool; females must be non-pregnant and not nursing.

Exclusion Criteria:

* Exclusion criteria include: diarrhea longer than 72 hours; moderate or severe dehydration, pregnancy or breast feeding, receipt of trimethoprim-sulfamethoxazole, azalide, doxycycline, or a fluoroquinolone in the past week; unstable medical condition; hypersensitivity to rifaximin or rifampin; fever (>100.6o F) or bloody diarrhea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316
Dates: Start 2004-06; Study Completion 2005-08

PRIMARY OUTCOMES:
The major outcome parameter was time from initiation of therapy until passage of the last unformed stool before becoming well (TLUS).

SECONDARY OUTCOMES:
Secondary Outcome Variables:
1. Time to passage of last unformed stool - standard definition of TLUS for antibiotics (18, 20) where wellness is declared at any time during 5 days regardless of later recurrence of continuing illness during the observation period;
2. Number of unformed stools passed during two days of therapy;
3. Number of unformed stools passed during the five days of study;
4. Improvement in diarrhea (<half the number of daily entry unformed stools in 24 hours) by 24 hours and 48 hours;
5. Treatment failure defined as: a. failure to achieve wellness during five days of study (achieve a TLUS-5 d); b. Deterioration during treatment and removed from further clinical evaluation, or, c. Occurrence of a relapse after achieving wellness during
6. Occurrence of relapse during five day surveillance (occurrence of diarrhea after having a TLUS);
7. TLUS in 48 hours - last unformed stool passed during the 48 hours that loperamide is being given (rapid symptomatic improvement);
8. Number of days of moderate or severe enteric symptoms;
9. Number of days passing any number of unformed stools plus any degree (mild, moderate or severe) of daily enteric symptoms (must have both present each day);
10. Subjects global assessment of efficacy by day of study;
11. Number of hours where schedule of activities were altered because of illness;
12. Number of hours confined to bed because of diarrhea;
13. Dropped from study due to adverse reaction;
14. Number of doses of loperamide (or loperamide placebos) taken;
15. Microbiologic eradication/failure.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert L. DuPont, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (4):
- Mexico (4):
  - Universidad Autonoma de Guadalajara, Guadalajara, Jalisco
  - University of Arizona, Colegio Guadalajara, Guadalajara, Jalisco
  - University of San Diego at Iteso, Guadalajara, Jalisco
  - Clinica Londres Morelos, Cuernavaca, Morelos